CLINICAL TRIAL: NCT06542458
Title: A Cohort Study of Older Adults From Under-resourced/Under-represented Communities Diagnosed With Subjective Cognitive Decline (SCD) or Mild Cognitive Disorder (MCI) Through Standard of Care Tele-Cog Visits (Tele-Cog)
Brief Title: Under-Represented Communities Diagnosed With SCD or MCI Through Tele-Cog
Status: Not yet recruiting | Type: Observational
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Douglas Scharre, Professor-Clinical, Ohio State University
Other Study IDs: NEW-64541
Record Dates: First submitted 2024-08-05; First posted 2024-08-07 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2024-08

CONDITIONS: Mild Cognitive Impairment; Subjective Cognitive Decline
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Study Population: Adults ages 50 years and older who are fluent in English and are diagnosed with subjective cognitive concerns (SCD) or objective cognitive decline with mostly intact functioning (MCI diagnosis) as part of clinical work up
  Interventions: Behavioral: Assessments; Other: Neuroimaging volumetric measures; Other: Biofluid samples

INTERVENTIONS:
Behavioral: Assessments — Participants will undergo a standard battery of neuropsychological measures, behavioral questionnaire, and functional assessment to monitor cognition and function over time. Clinical data obtained as part of standard of care will be collected from the medical record
Other: Neuroimaging volumetric measures — Neuroimaging volumetric measures will be obtained from already conducted standard of care neuroimaging.
Other: Biofluid samples — Biofluid sampling data will be obtained through another protocol. All participants will be required to sign that consent to participate in this trial.

SUMMARY:
Overall, this study's primary aim is to establish a prospective, longitudinal, observational cohort study of older adults at risk for dementia from under-resourced/underrepresented communities. More specifically, older adults diagnosed with subjective cognitive decline (SCD) or Mild Cognitive Impairment (MCI) during clinical care offered via the Tele-Cog clinic would be recruited for more comprehensive data collection to characterize the clinical presentation and course of illness over multiple timepoints spread out longitudinally.

DETAILED DESCRIPTION:
Clinical data obtained as part of standard of care will be collected from the medical record (including clinical diagnosis, cognitive and other neuropsychological test scores, lab results, neuroimaging data, etc.) and additional data (neuropsychological test batteries and clinical questionnaires if not already obtained) would be obtained at research study visits.

Participants will be asked to participate in annual research visits for up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

1. Adults ages 50 years and older
2. Diagnosed with subjective cognitive concerns (SCD) or objective cognitive decline with mostly intact functioning (MCI diagnosis) as part of clinical work up
3. Fluent in English
4. Able to provide voluntary informed consent
5. Willing and able to undergo all study procedures
6. Able to delegate, if possible, a study partner to contribute information regarding daily activities and cognition

Exclusion Criteria:

1. Diagnosis of dementia at baseline.
2. Inability to give informed consent.
3. High risk of adverse emotional or behavioral reaction based on investigator's clinical evaluation (e.g., evidence of serious personality disorder, antisocial behavior, serious current stressors, lack of meaningful social support).

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals will be recruited from the Tele-Cog clinic at The Ohio State University Wexner Medical Center.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2032-01-01 (Estimated); Study Completion 2032-01-01 (Estimated)

PRIMARY OUTCOMES:
Number of adults with Subjective Cognitive Decline (SCD) or Mild Cognitive Impairment (MCI) at risk for dementia from under-resourced/underrepresented communities that we longitudinally collect clinical data, neuropsychology, neuroimaging, and biofluids | 5 years
  This study is a longitudinal collection of clinical data, neuroimaging, neuropsychological assessments, and biofluids to establish a cohort of older adults with Subjective Cognitive Decline (SCD) or Mild Cognitive Impairment (MCI) at risk for dementia from under-resourced/underrepresented communities from which hypotheses can be generated. Analysis will also include comparing the subject's longitudinal change over time data. Data will be analyzed with one way and repeated measures (ANOVAs) that will control for important covariates. All imaging data will be analyzed using qualitative visual interpretation and quantitative region of interest approach.

CONTACTS AND LOCATIONS:
Locations (1):
- The Ohio State University, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No